CLINICAL TRIAL: NCT01016067
Title: A Prospective, Randomized, Multicenter Pivotal Clinical Trial of the INFUSE/MASTERGRAFT™ Delayed Healing Device With Rigid Internal Fixation in the Treatment of Tibial Delayed Healing
Brief Title: Tibial Delayed Healing Pivotal Clinical Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in patient recruitment
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Medtronic P07-01
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Tibial Delayed Healing
Keywords: Tibia; Tibial; Fracture; Nonunion; delayed; healing; iliac; crest; autograft; INFUSE; MASTERGRAFT; Fixation; Internal
MeSH Terms: conditions — Fractures, Bone; Scleroderma, Limited

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INFUSE/MASTERGRAFT (Experimental): Patients received INFUSE/MASTERGRAFT granules with rigid internal fixation.
  Interventions: Device: INFUSE/MASTERGRAFT
- Autograft bone (Active Comparator): Patients received autograft bone with rigid internal fixation.
  Interventions: Procedure: Autograft bone

INTERVENTIONS:
Device: INFUSE/MASTERGRAFT — INFUSE® (rhBMP-2) on an absorbable collagen sponge (ACS) and MASTERGRAFT® granules with appropriate rigid internal fixation hardware (reamed IM nail or plate/screws)
  Other Names: INFUSE; MASTERGRAFT
  Arms: INFUSE/MASTERGRAFT
Procedure: Autograft bone — Autogenous bone graft with appropriate rigid internal fixation hardware (reamed IM nail or plate/screws)
  Other Names: Autogenous bone graft
  Arms: Autograft bone

SUMMARY:
Evaluate the INFUSE/MASTERGRAFT™ Delayed Healing Device as an alternative/replacement to autograft in the treatment of tibial delayed healing.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the INFUSE/MASTERGRAFT™ Delayed Healing Device as an alternative/replacement to autograft in the treatment of tibial delayed healing. A subject will be considered to have tibial delayed healing when he/she is at least six months from the date of the most recent surgical intervention and has shown no signs of radiographic healing for at least three months. Radiographic signs of healing for this study are defined as either the progressive disappearance of fracture lines or the development of cortical continuity [bridging bone] at the site. All prospective patients must require surgical treatment with rigid internal fixation [reamed IM nail or plate/screws] and bone grafting.

ELIGIBILITY:
Inclusion Criteria:

1. Has tibial delayed healing. A subject will be considered to have delayed healing when he/she is at least six months from the date of the most recent surgical intervention and has shown no signs of radiographic healing for at least three months. (Radiographic signs of healing for this study are defined as either the progressive disappearance of fracture lines or the development of cortical continuity [bridging bone] at the site.)
2. Has delayed healing of the tibia that requires treatment with rigid internal fixation and bone grafting. (Stable rigid internal fixation hardware may already be in place prior to treatment. If required, the fixation hardware may be removed and replaced along with the placement of the bone graft.)
3. Has adequate soft tissue coverage at the delayed healing site. All prior soft tissue coverage procedures (e.g., skin grafts or flaps) should be sufficiently healed for placement of a bone graft prior to enrollment in the study.
4. Has a sufficient amount of iliac crest autograft available for a bone grafting procedure.
5. After walking 5 or 6 steps, has intensity of pain/discomfort at the injury site equal to or greater than 4 (as reported on the preoperative Delayed Healing Site Pain Questionnaire form; 0 being no pain and 10 being pain as bad as it could be).
6. Is at least 21 years of age and skeletally mature at the time of surgery.
7. If a female of child-bearing potential, patient is not pregnant or nursing and agrees not to become pregnant for one year following surgery in the study.
8. Is willing and able to comply with the study plan and able to understand and sign the Patient Informed Consent Form.

Exclusion Criteria:

1. Has a congenital pseudarthrosis or pathological fracture nonunion (not including osteoporosis-related fractures).
2. Has a tibial delayed healing with articular involvement (e.g., intra-articular). (The original fracture may have involved the joint, but the resulting delayed healing site may not involve the joint.)
3. Has hypertrophic tibial delayed healing (e.g., observed on x-ray as having an abundant callus or "horse hoof" appearance).
4. Has inadequate neurovascular status in the involved limb that may jeopardize healing.
5. Has an active or a known prior infection at the delayed healing site (e.g., the presence of purulent drainage from the site, prior positive cultures from the site, or evidence of active/prior osteomyelitis at the site). Enrolled subjects whose intra-operative cultures test positive for bacteria may remain in the study.
6. Has existing stable hardware that will not be removed and does not meet the algorithm requirements.
7. Has treatment planned for the delayed healing that does NOT include placement of a bone graft and/or rigid internal fixation consisting of a reamed intramedullary nail or plate/screws.
8. Has a tibial delayed healing injury site with a bony defect larger than 4 cm in length.
9. Has another injury/condition that prevents ambulation or completion of any of the study assessments.
10. Has a history of endocrine or metabolic disorder known to affect osteogenesis (e.g., Paget's disease, renal osteodystrophy, hyperthyroidism, parathyroid hormone disorder, Ehler-Danlos syndrome, osteogenesis imperfecta, calcium imbalance).
11. Has a Vitamin D deficiency, defined as a 25-hydroxy Vitamin D serum concentration of ≤11ng/mL .
12. Has an active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
13. Has an overt or active systemic infection (e.g., HIV/AIDS, hepatitis, bacteremia).
14. Has been on oral or injectable steroids for six weeks or more at time of enrollment. This does not include episodic steroid use; inhaled steroids; or steroid medication (e.g., Epidural Steroid Injections, Medrol DosePaks) specifically for the perioperative management of symptoms.
15. Has a condition requiring postoperative medications that could interfere with bone healing of the implant, such as steroids. This does not include low dose aspirin for prophylactic anticoagulation; routine perioperative anti-inflammatory drugs; episodic steroid use; or inhaled steroids.
16. Has a history of certain autoimmune diseases. (Refer to the List of Autoimmune Diseases in the CIP for further information.)
17. Has a history of exposure to injectable collagen or silicone implants.
18. Has any previous exposure to any recombinant BMPs of either human or animal extraction.
19. Has a history of hypersensitivity to collagen or protein pharmaceuticals (e.g., monoclonal antibodies or gamma globulins).
20. Has a history of allergy to bovine collagen products.
21. Has a documented allergy or intolerance to metal or metal alloys, such as stainless steel or titanium.
22. Has chronic or acute renal and/or hepatic failure or prior history of renal and/or hepatic parenchymal disease.
23. Is mentally incompetent. If questionable, obtain psychiatric consult.
24. Is a prisoner.
25. Is an alcohol and/or drug abuser as defined by currently undergoing treatment for alcohol and/or drug abuse.
26. Has received treatment with an investigational therapy (drug, device, and/or biologic) within 28 days prior to implantation surgery or such treatment is planned during the 12-month period following the study surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Denver Health, Denver, Colorado
  - Shrock Orthopedic Research, Fort Lauderdale, Florida
  - University of Florida College of Medicine, Jacksonville, Florida
  - Orlando Health, Orlando, Florida
  - Fort Wayne Orthopaedics, Fort Wayne, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Missouri, Columbia, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Lutheran Medical Center, Brooklyn, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Ohio Health Research Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Geisinger Clinic, Danville, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Started | 11 | 12
Completed | 9 | 8
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrew due to Relocation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.76) | 37.7 (8.47) | 42.5 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 11 | 8 | 19
  Black | 0 | 4 | 4
  Asian | 0 | 0 | 0
  Hispanic | 0 | 0 | 0
  Other | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: Inches] | 69.0 (3.44) | 68.6 (4.56) | 68.8 (3.98)
Weight [Mean (Standard Deviation); unit: lbs.] | 178.9 (50.07) | 186.3 (42.74) | 182.7 (45.46)

OUTCOME MEASURES:

1. Primary Outcome: Overall Success
Description: Overall success is reported as participants who met all of the following criteria: 1. radiographic union success; 2. success in weight bearing ability; 3. improvement in pain at the delayed healing site; 4. no serious adverse event classified as "implant-associated" or "implant/surgical procedure-associated" (device-related); 5.no additional surgical procedures classified as a failure.
Time Frame: 12 Months
Population: Ten investigational and 9 control subjects were evaluable for overall success while only 9 investigational and 8 control subjects completed the study at 12-month follow-up. Two subjects were classified as "failure" due to related serious adverse event or additional surgery before completion of the study.
Measure: Number; unit: participants
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Number analyzed (Participants) | 10 | 9
participants | 7 | 1

2. Secondary Outcome: Radiographic Union Success
Description: Radiographic union success (a component of overall success) was defined as complete disappearance of fracture lines or the presence of bridging bone across the delayed healing site as observed on at least three of the four cortices (anterior, posterior, medial, and lateral), using plain films. If there was more than one delayed healing fracture line, all fracture lines must have been united in order to be considered a successful fracture union.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Number analyzed (Participants) | 9 | 8
participants | 9 | 6

3. Secondary Outcome: Success in Weight Bearing Ability
Description: Success in weight bearing ability (a component of overall success) was defined that subject was able to bear weight without severe pain on the affected limb. The subject was asked to stand, bearing full weight on the affected limb in a single-leg stance without ambulatory assistance for 10 seconds. If the subject was able to do so without severe pain, a positive (success) response was recorded. If the subject was either unable to stand on the affected limb in a single-leg stance or declined to do so because of limb weakness, poor balance, or severe leg pain, a negative (failure) response was documented.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Number analyzed (Participants) | 9 | 8
participants | 9 | 7

4. Secondary Outcome: Success of Pain Status at the Delayed Healing Site
Description: After walking five or six steps, subjects rated their intensity of pain/discomfort at the delayed healing site using a numerical rating scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be". Subjects who were unable or declined to walk because of severe leg pain were considered to have a score of 10. Success for pain at the delayed healing site was defined as at least a 2-point improvement in pain from the pre-operative score. Success of pain status at the delayed healing site was a component of overall success.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Number analyzed (Participants) | 9 | 8
participants | 7 | 3

5. Secondary Outcome: Success in Short Musculoskeletal Functional Assessment (SMFA)
Description: The SMFA is an assessment tool that measures a subject's overall function for a broad range of musculoskeletal injuries and disorders. The SMFA results were summarized into two components, the dysfunctional index and the bother index. Success for the SMFA assessment was defined as any improvement post-operatively as compared to the pre-operative condition.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Number analyzed (Participants) | 9 | 8
participants
  SMFA Dysfunctional Index Success | 7 | 8
  SMFA Bother Index Success | 6 | 6

6. Secondary Outcome: Success in Short Form 36-Item (SF-36) Health Survey
Description: SF-36 was used to assess general health status. The SF-36 results were summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). Success was defined as any improvement in a subject's SF-36 PCS post-operatively as compared to the pre-operative condition.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Number analyzed (Participants) | 9 | 8
participants | 8 | 7

7. Secondary Outcome: Number of Subjects Having Additional Surgical Procedure Classified as a Treatment "Failure"
Description: Subject who had a surgery after the original study treatment was classified as a treatment "failure" if the additional surgery or treatment occurred in the involved limb and affected the study treatment and/or its mechanism of action in relation to the diagnosis or condition of the subject that was the cause for having the original study treatment.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Number analyzed (Participants) | 11 | 12
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: All study periods
Arm/Group | INFUSE/MASTERGRAFT | Autograft Bone
Serious Adverse Events (participants affected / at risk) | 5/11 | 3/12
Other Adverse Events (participants affected / at risk) | 7/11 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFUSE/MASTERGRAFT (N=11) | Autograft Bone (N=12)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Completed Suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFUSE/MASTERGRAFT (N=11) | Autograft Bone (N=12)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Device component issue (General disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Medical device discomfort (General disorders) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemoglobin decresed (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was terminated due to difficulty in patient recruitment. Early termination led to a small number of subjects analyzed. Results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less